CLINICAL TRIAL: NCT06534268
Title: Study on Postoperative Adrenal Function Assessment in Patients With Primary Aldosteronism
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RJ-PA-NEW-1
Record Dates: First submitted 2024-07-27; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — patient serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study employs a prospective, single-center, open, observational research design to evaluate postoperative adrenal cortical function in patients with primary aldosteronism (PA) and to explore indicators predicting postoperative adrenal insufficiency and their predictive efficacy

DETAILED DESCRIPTION:
Patients suspected of having primary aldosteronism and admitted for treatment, who are diagnosed with primary aldosteronism through at least one confirmatory test, and subsequently diagnosed with unilateral primary aldosteronism via bilateral adrenal vein sampling and ACTH stimulation test, will undergo surgery. Those who have an ACTH stimulation test within one week postoperatively will be included in the study.

This study employs a prospective, single-center, open, observational research design to evaluate postoperative adrenal cortical function in patients with primary aldosteronism (PA) and to explore indicators predicting postoperative adrenal insufficiency and their predictive efficacy

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unilateral primary aldosteronism who undergo surgical treatment and have their cortical function assessed by an ACTH stimulation test within one week postoperatively.

Exclusion Criteria:

* Patients using medications that affect adrenal cortical function.
* Patients with a history of adrenal surgery
* Pregnant or breastfeeding women
* Patients with severe underlying diseases (such as liver or kidney failure) that may affect adrenal cortical function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study intends to include 200 patients diagnosed with primary aldosteronism undergoing surgery. An ACTH stimulation test will be performed within one week postoperatively. The participants will be aged 18-75 years, with no gender restrictions. Exclusion criteria include patients using medications that affect adrenal cortical function, patients with a history of adrenal surgery, pregnant or breastfeeding women, and patients with severe underlying diseases (such as liver or kidney failure) that may affect adrenal cortical function
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The gender and age of the participants | 1 day
  age in years and sex (female or male) of patients
Participant's weight and height | 1 day
  BMI(body mess index) in kg/m^2= (weight in kg) /(height in m)^2
Patients' baseline hormone level | 1day
  serum hormone level
Number of Participants with baseline glucose metabolic levels | 1 day
  glucose metabolism, lipid metabolism, liver and kidney function, electrolytes, etc
Patients' hormone levels at 0 minutes and 120 minutes after preoperative ACTH stimulation test | 1day
  cortisol and aldosterone levels
Patients' hormone levels at 0 minutes and 120 minutes after postoperative ACTH stimulation test | 1day
  cortisol and aldosterone levels
Number of Participants with baseline lipid metabolic levels | 1day
  blood lipid levels
Patients' baseline glucose metabolic levels | 1day
  0-minute、30-minute、60-minute 、120-minute and 180-minute blood glucose levels after OGTT
Number of Participants with baseline electrolytes levels | 1day
  sodium, potassium, chloride, calcium, and phosphorus ion levels
Number of Participants with baseline kidney function levels | 1day
  Creatinine, blood urea nitrogen (BUN), and uric acid levels

SECONDARY OUTCOMES:
the changes of hormone levels after surgical management | 1day
  cortisol and aldosterone serum hormone level
Number of Participants with changes of lipid metabolic levels after surgical management | 1day
  blood lipid levels
the changes of glucose metabolic levels after surgical management | 1day
  0-minute、30-minute、60-minute 、120-minute and 180-minute blood glucose levels after OGTT
Number of Participants with changes of kidney function levels after surgical management | 1 day
  Creatinine, blood urea nitrogen (BUN), and uric acid levels

IPD SHARING:
Plan to Share IPD: Yes